CLINICAL TRIAL: NCT03771729
Title: Observation on the Effect of Sacubitril/Valsartan in Advanced Chronic Kidney Disease（CKD）Patients With Heart Failure
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Xuanyi Du, Principal Investigator, The Second Affiliated Hospital of Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42411671-X
Record Dates: First submitted 2018-11-30; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: CKD
Keywords: Sacubitril/Valsartan; Advanced CKD Patients; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCZ696 treatment (Experimental): LCZ696 200mg twice daily
  Interventions: Drug: LCZ 696

INTERVENTIONS:
Drug: LCZ 696 — LCZ696 200mg twice daily
  Other Names: sacubitril/valsartan

SUMMARY:
This paper will mainly present the renal results from a clinical study aimed to observe the effect of sacubitril/valsartan in advanced chronic kedney disease patients with heart failure.All patients will receive LCZ696.The results will be compared before and after treatment.

DETAILED DESCRIPTION:
On trial entry, patients will first receive LCZ696 50mg twice daily.According to the condition of disease and tolerance,the dose will be doubled every 2 weeks until the target maintenance dose 200mg twice daily is reached unless potassium or change in kidney function preclude a dose increase(reduction in dose will be permitted if the larger dose will not be tolerated, and temporary interruption will be permitted at any time if required for clinical reasons).The trial will be followed up for 12 weeks. Study visits will be scheduled at 2,4,6,8,10and12 weeks (and additional visits will be arranged where necessary to monitor participant safety).

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with Chronic kidney disease (eGFR<60 ml/ min/1.73m²) and heart failure
2. documented history of heart failure with associated signs or symptoms
3. New York Heart Association (NYHA) classes II-IV
4. mean sitting systolic blood pressure (msSBP) ⩾140mmHg
5. good compliance

Exclusion Criteria:

1. isolated right heart failure owing to pulmonary disease, dyspnoea from non-cardiac causes, primary valvular or myocardial diseases, or coronary or cerebrovascular diseases needing revascularization within 3months of screening or during the trial
2. acute renal failure
3. systolic blood pressure lower than 100 mm Hg at screening (<95 mm Hg at the randomisation visit)
4. significant laboratory abnormalities at screening interfering with assessment of study drug safety or efficacy(such as serum potassium>5.5 or <3.5mmol/L, serum sodium<130mmol/L or alanine aminotransferase or aspartate aminotransferase>2 times the upper limit of the normal range)
5. history of angioedema（drug-related or otherwise)
6. any medications that have potential for drug-drug interaction with LCZ696 will not be allowed during the study 7)pregnant female

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-30 (Estimated); Primary Completion 2019-05-28 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate(eGFR) | 12 weeks
  Blood samples will be collected for analysis of glomerular filtration rate(eGFR) every 2weeks .
Change in urinary microalbumin/creatinine ratio(uACR) | 12 weeks
  Urine samples will be collected for analysis of urinary microalbumin/creatinine ratio(uACR) every 2weeks.
Concentration of N terminal pro B type natriuretic peptide(NT-prpBNP) | 12 weeks
  Blood samples will be collected for analysis of concentration of N terminal pro B type natriuretic peptide(NT-proBNP) every 2weeks.

SECONDARY OUTCOMES:
blood uric acid | 12 weeks
  Blood samples will be collected for analysis of uric acid every 2weeks.
Rate of HbA1c | 12weeks
  Blood samples will be collected for analysis of HbA1c every 2weeks.
Systolic and diastolic blood pressure | 12 weeks
  Systolic and diastolic blood pressure will be measured every 2weeks.
left ventricle eject fraction | 12 weeks
  Cardiac ultrasound will be measured every 2weeks.
Concentration of postassium | 12 weeks
  Blood samples will be collected for analysis of concentration of postassium every 2weeks.
Concentration of serum troponin | 12 weeks
  Blood samples will be collected for analysis of concentration of serum troponin every 2weeks.
Concentration of alanine aminotransferase or aspartate aminotransferase | 12 weeks
  Blood samples will be collected for analysis of concentration of alanine aminotransferase or aspartate aminotransferase every 2weeks.
Concentration of sodio | 12 weeks
  Urine samples will be collected for analysis of concentration of sodion every 2weeks.

IPD SHARING:
Plan to Share IPD: Undecided
Clinical Study Report (CSR)